CLINICAL TRIAL: NCT02010944
Title: An Open-label, Parallel Group, Randomized, Two-sequence, Three-way Crossover Study to Assess the Relative Bioavailability of Solifenacin Succinate and Mirabegron Fixed-dose Combination Tablets Compared to Co-administration of Single Entity Tablets at Three Dose Strengths in Healthy Male and Female Subjects
Brief Title: A Study to Compare How Much Solifenacin Succinate and Mirabegron Reach the Blood When Administered Together as Fixed-dose Combination Tablets and With Single Individual Tablets of the Same Medications at Three Dose Levels
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Europe B.V. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 178-CL-103; 2012-002650-23 (EudraCT Number)
Record Dates: First submitted 2013-10-04; First posted 2013-12-13 (Estimated); Last update posted 2013-12-13 (Estimated); Status verified 2013-10

CONDITIONS: Phase 1; Bioavailability; Healthy Subjects
Keywords: Solifenacin; Mirabegron; Fixed-dose combination (FDC); Single Entity Tablet (SET); Pharmacokinetics; Bioavailability
MeSH Terms: interventions — Solifenacin Succinate; mirabegron

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1: FDC-SET-SET (Experimental): Fixed Dose Combination followed by two periods of the Single Entity Tablets
  Interventions: Drug: solifenacin succinate; Drug: mirabegron; Drug: mirabegron/solifenacin succinate
- 2: SET-FDC-FDC (Experimental): Single Entity Tablets followed by two periods of Fixed Dose Combination
  Interventions: Drug: solifenacin succinate; Drug: mirabegron; Drug: mirabegron/solifenacin succinate

INTERVENTIONS:
Drug: solifenacin succinate — oral
  Other Names: Vesicare®,; YM905
Drug: mirabegron — oral
  Other Names: YM178
Drug: mirabegron/solifenacin succinate — oral
  Other Names: YM178/YM905

SUMMARY:
This study compares the pharmacokinetics (PK), safety and tolerability of fixed dose combination (FDC) tablets containing solifenacin succinate and mirabegron with the co-administration of single entity tablets (SET), at three dose strengths.

DETAILED DESCRIPTION:
There are three parallel groups each with 24 healthy male and female subjects (with a minimum of 10 subjects per gender). Each group receives one dose strength.

The study utilizes a partial replicate cross-over design with three periods and each subject receives the same strength of either the FDC or SET formulation twice.

Screening takes place within 21 days before admission and subjects are admitted on Day -1. Dosing takes place on Day 1, after an overnight fast of at least 10 hours. Subjects remain fasted until 4 hours post-dose. There is a wash-out period of at least 14 days between each dose administration.

Subjects are discharged on Day 4 and return to the clinical unit on Days 5, 6, 7, 9 and 11 for outpatient assessments.

An End-of-Study Visit (ESV) takes place on Day 11 of Period 3 or within 7-14 days after discontinuation.

ELIGIBILITY:
Inclusion Criteria:

* Male subject must agree to not donate semen from the day of first dosing until 3 months after last discharge and practice an effective contraceptive method with female sexual partners to prevent pregnancy.
* Female subject must be of non-child bearing potential, i.e. postmenopausal, surgically sterilized, hysterectomy in medical history, or practicing highly effective non-hormonal birth control.

Exclusion Criteria:

* Female subject who is pregnant, has been pregnant within 6 months before screening or breast-feeding within 3 months before screening.
* Known or suspected hypersensitivity to solifenacin succinate, mirabegron or any components of the formulations used.
* The subject has/had febrile illness or symptomatic, viral, bacterial (including upper respiratory infection), or fungal (non-cutaneous) infection within 1 week prior to admission to the clinical unit.
* Any significant blood loss, donated one unit (450 mL) of blood or more, or received a transfusion of any blood or blood products within 60 days or donated plasma within 7 days prior to clinic admission on Day -1.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2012-09; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic parameter of solifenacin in plasma as measured by Cmax (Maximum concentration) | Days 1-11
Pharmacokinetic parameter of solifenacin in plasma as measured by AUClast (AUC until last sample taken) | Days 1-11
Pharmacokinetic parameter of solifenacin in plasma as measured by AUCinf (AUC extrapolated until infinity) | Days 1-11
Pharmacokinetic parameter of mirabegron in plasma as measured by Cmax (Maximum concentration) | Days 1-11
Pharmacokinetic parameter of mirabegron in plasma as measured by AUClast (AUC until last sample taken) | Days 1-11
Pharmacokinetic parameter of mirabegron in plasma as measured by AUCinf (AUC extrapolated until infinity) | Days 1-11

SECONDARY OUTCOMES:
Pharmacokinetic profile of Solifenacin in plasma | Days 1-11
  AUC0-72h (Area under the plasma concentration-time curve from time zero to 72h), tmax (Time to attain Cmax), tlag (Absorption lag time), t1/2 (Apparent terminal elimination half-life), Vz/F (Apparent volume of distribution), CL/F (Apparent total body plasma clearance)
Pharmacokinetic profile of mirabegron in plasma | Days 1-11
  AUC0-72h (Area under the plasma concentration-time curve from time zero to 72h), tmax (Time to attain Cmax), tlag (Absorption lag time), t1/2 (Apparent terminal elimination half-life), Vz/F (Apparent volume of distribution), CL/F (Apparent total body plasma clearance)
Safety and tolerability of solifenacin succinate and mirabegron assessed by adverse events, vital signs, laboratory tests, physical examination and 12-lead electrocardiogram (ECG) | Screening to End of Study Visit (Day 11 Period 3 or within 7 to 14 days after discontinuation)

CONTACTS AND LOCATIONS:
Overall Officials: Study Manager, Study Chair — Astellas Pharma Europe B.V.
Locations (1):
- Parexel, Berlin, Germany